CLINICAL TRIAL: NCT01038427
Title: A Double-Blind, Randomized, Placebo Controlled, Parallel Group, Multi-Site Study to Compare the Clinical Equivalence of Mometasone Nasal Spray (Lek Pharmaceuticals) With NASONEX® Nasal Spray (Schering Corporation) in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Brief Title: A Study Comparing the Clinical Equivalence of Two Mometasone Nasal Sprays in the Relief of the Signs and Symptoms of Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70947201
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Rhinitis; Seasonal Allergic Rhinitis; Mometasone Furoate; Equivalence; Hay fever
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Test (Experimental): Mometasone furoate 50 mcg/actuation nasal spray (Lek Pharmaceuticals) administered once daily at a dose of 200 mcg (4 actuations) for 14 days.
  Interventions: Drug: Mometasone furoate 50 mcg/actuation nasal spray (Lek Pharmaceuticals)
- Reference (Active Comparator): Mometasone furoate (Nasonex®) 50 mcg/actuation nasal spray administered once daily at a dose of 200 mcg (4 actuations) for 14 days.
  Interventions: Drug: Mometasone furoate (Nasonex®) 50 mcg/actuation nasal spray
- Placebo (Placebo Comparator): Placebo nasal spray administered once daily for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate 50 mcg/actuation nasal spray (Lek Pharmaceuticals) — Mometasone nasal spray administered once daily at a dose of 200 mcg (4 actuations) for 14 days.
  Arms: Test
Drug: Mometasone furoate (Nasonex®) 50 mcg/actuation nasal spray — Mometasone nasal spray administered once daily at a dose of 200 mcg (4 actuations) for 14 days.
  Arms: Reference
Drug: Placebo — Placebo nasal spray administered once daily (4 actuations) for 14 days.
  Arms: Placebo

SUMMARY:
This study compared the efficacy and safety of a generic mometasone nasal spray to the reference listed drug in the treatment of seasonal allergic rhinitis. Additionally both the test and the reference formulations were tested for superiority against a placebo nasal spray.

DETAILED DESCRIPTION:
The study was designed as a double-blind, randomized, placebo-controlled, parallel group, multi-site to compare the clinical equivalence of the test formulation of mometasone furoate monohydrate, 50 mcg/actuation nasal spray (Lek Pharmaceuticals d.d.) with the reference formulation Nasonex® nasal spray (Schering) in the relief of the signs and symptoms of seasonal allergic rhinitis. Participants who met the inclusion/exclusion criteria entered a 7-day placebo lead-in period. Following this placebo lead-in period, on Day 1 participants who continued to meet eligibility criteria were randomly assigned in a 2:2:1 ratio to one of three treatment groups (Test Product:Reference Product:Placebo) for 14 days of treatment. In all treatment groups, participants were instructed to administer the study drug once daily at approximately the same time each day. A single dose of 200 mcg was 4 actuations, each containing 50 mcg per actuation. Patients were instructed to administer the 4 actuations alternating between right and left nostril, such that 2 actuations were not administered back to back to the same nostril.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female 12 years of age or older with a minimum of 2 years of previous history of seasonal allergic rhinitis to the pollen/allergen in season at the time the study is being conducted.
* Signed informed consent form. For patients under the age of majority the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form.
* Documented positive allergic skin test to local pollen, performed within the past 12 months.
* A score of at least 6 on the reflective Total Nasal Symptom Score (rTNSS) with a minimum score of at least 2 for "nasal congestion" and a minimum score of at least 2 for one of the remaining 3 symptoms.

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.
* History of asthma over the previous two years that required chronic therapy (with the exception of occasional acute or mild exercise induced asthma).
* Patients with some nasal conditions, or with clinically significant nasal deformity or any recent nasal surgery or trauma that has not completely healed.
* Upper respiratory tract infection or any untreated infections within the previous 30 days.
* Patient has started immunotherapy/changed the dose within 30 days of starting the study or has desensitization therapy to the seasonal allergen that is causing the allergic rhinitis within the previous 6 months.
* Patients with a history of tuberculosis, or with the presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis or other eye infection not related to the diagnosis of seasonal allergic rhinitis within 14 days of enrollment.
* The patient has had recent exposure (30 days) or was at risk of being exposed to chicken pox or measles.
* Any known hypersensitivity to mometasone, other steroids or any of the components of the study nasal spray.
* Planned travel outside of the local area for more than 2 consecutive days or 3 days in total.
* The patient has a history of alcohol or drug abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 795 (Actual)
Dates: Start 2009-12-02 (Actual); Primary Completion 2010-02-16 (Actual); Study Completion 2010-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Austin, Texas
  - Kerrville, Texas
  - Live Oak, Texas
  - New Braunfels, Texas
  - Sylvana Research, San Antonio, Texas
  - San Antonio, Texas
  - Waco, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 10 investigative sites in 1 country.
Pre-assignment Details: Participants who met the inclusion/exclusion criteria entered a 7-day placebo lead-in period. Following this placebo lead-in period, on Day 1 participants who continued to meet eligibility criteria were randomly assigned in a 2:2:1 ratio to one of three treatment groups (Test Product:Reference Product:Placebo).
Period: Overall Study
Arm/Group | Test | Reference | Placebo
Started | 317 | 320 | 158
Per-Protocol (PPP) Population (All participants who satisfied the criteria set forth in the protocol in terms of dosing compliance, number of available post-randomization evaluations and absence of significant protocol violations.) | 306 | 307 | 150
Intent-to-Treat (ITT) Population (All participants in the PPP as well as all participants who administered at least one dose of randomized study drug and had at least one post-randomization evaluation.) | 314 | 314 | 156
Completed | 314 | 314 | 154
Not Completed | 3 | 6 | 4
Not completed — Lost to follow up | 1 | 1 | 0
Not completed — Restricted medication for seasonal allergic rhinitis | 0 | 0 | 1
Not completed — Withdrew consent | 0 | 0 | 1
Not completed — Adverse Event | 2 | 2 | 1
Not completed — Enrolled in error | 0 | 1 | 1
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Reference | Placebo | Total
Number analyzed (Participants) | 317 | 320 | 158 | 795
Age, Customized [Count of Participants; unit: Participants]
  < 18 | 28 | 39 | 12 | 79
  18 - 40 | 147 | 139 | 77 | 363
  41 - 64 | 130 | 125 | 63 | 318
  65 - 75 | 9 | 16 | 5 | 30
  > 75 | 3 | 1 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 205 | 207 | 109 | 521
  Male | 112 | 113 | 49 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 271 | 277 | 140 | 688
  Black/African American | 39 | 35 | 15 | 89
  Asian | 4 | 2 | 1 | 7
  Native Hawaiian / Other Pacific Islander | 1 | 1 | 1 | 3
  Other | 2 | 5 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Reflective Total Nasal Symptom Score (rTNSS) (Equivalence: Per-Protocol Population)
Description: Patients were required to record a 12 hour "reflective" score twice a day approximately 12 hours apart. For the rTNSS patients were asked to "look back" or "reflect" on their severity of nasal symptoms over the previous 12 hours. The first rating on each day was taken prior to dosing. Patients were asked to score 4 nasal symptoms (nasal congestion, runny nose, sneezing and itchy nose) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 4 individual symptom scores obtained over the randomized treatment period were summed to give the mean rTNSS, which ranged from 0 to 12 with a lower score indicating less severe symptoms.
  Mean baseline rTNSS was calculated by summing the means of the 4 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline rTNSS" - "mean post-randomization rTNSS". A positive change from baseline in rTNSS is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: Per-Protocol population was used in this analysis. To determine equivalence, only the test and reference treatment arms were analyzed.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 306 | 307
score on scale | 1.981 (2.335) | 1.817 (2.258)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — If the 90% confidence intervals were contained within the interval 80.0% to 125.0%, then the two products were considered to be therapeutically equivalent; Ratio Test/Ref. Least Squares (LS) Means = 106.644, 90% CI 2-sided [91.860 to 123.997]

2. Primary Outcome: Mean Change From Baseline in Reflective Total Nasal Symptom Score (rTNSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 1
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 311 | 311 | 153
score on scale | 2.008 (2.356) | 1.794 (2.257) | 1.034 (1.894)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0001, ANCOVA

3. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (iTNSS) (Equivalence: Per-Protocol Population)
Description: Patients were required to record an "instantaneous" score twice a day approximately 12 hours apart. For the iTNSS patients were asked to evaluate "how I feel now" regarding their severity of nasal symptoms. The first rating on each day was taken prior to dosing. Patients were asked to score 4 nasal symptoms (nasal congestion, runny nose, sneezing and itchy nose) on a 4 point scale ranging from 0 (no symptom) to 3 (severe symptom). The means of the 4 individual symptom scores obtained over the randomized treatment period were summed to give the mean iTNSS, which ranged from 0 to 12 with a lower score indicating less severe symptoms.
  Mean baseline iTNSS was calculated by summing the means of the 4 individual symptom scores obtained over the 72 hours before the randomized treatment period.
  Mean change from baseline was calculated as "mean baseline iTNSS" - "mean post-randomization iTNSS". A positive change from baseline in iTNSS is considered a favorable outcome.
Time Frame: Baseline, 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference
Number analyzed (Participants) | 306 | 307
score on scale | 1.900 (2.408) | 1.656 (2.207)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — 90% confidence intervals within the interval 80.0% to 125.0%; Ratio Test/Ref. LS Means = 109.716, 90% CI 2-sided [93.316 to 129.159]

4. Secondary Outcome: Mean Change From Baseline in Instantaneous Total Nasal Symptom Score (iTNSS) (Superiority: Intent-to-Treat Population)
Description: as for outcome 3
Time Frame: Baseline, 14 days
Population: Intent-to-Treat Population including participants with valid measurements for the outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 311 | 311 | 153
score on scale | 1.932 (2.419) | 1.630 (2.214) | 0.905 (1.914)
Statistical Analysis 1: Comparison: Test vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Reference vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

5. Secondary Outcome: Clinical Global Improvement Based on the Investigator's Assessment
Description: A global evaluation of efficacy relative to baseline was assessed separately by the investigator and the patient on Day 15. Both the investigator and the patient were asked to rate clinical improvement since baseline on a 5-category scale ranging from "No Relief" to "Complete Relief" of signs and symptoms of seasonal allergic rhinitis. This record shows the clinical global improvement based on the investigator's assessment.
Time Frame: Day 15
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 314 | 314 | 156
Participants
  No Relief | 34 | 53 | 39
  Slight Relief | 83 | 72 | 38
  Moderate Relief | 125 | 119 | 56
  Marked Relief | 68 | 67 | 23
  Complete Relief | 4 | 3 | 0
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Superiority; p = 0.2655, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.1093, Cochran-Mantel-Haenszel

6. Secondary Outcome: Clinical Global Improvement Based on the Patient's Assessment
Description: A global evaluation of efficacy relative to baseline was assessed separately by the investigator and the patient on Day 15. Both the investigator and the patient were asked to rate clinical improvement since baseline on a 5-category scale ranging from "No Relief" to "Complete Relief" of signs and symptoms of seasonal allergic rhinitis. This record shows the clinical global improvement based on the patient's assessment.
Time Frame: Day 15
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference | Placebo
Number analyzed (Participants) | 314 | 314 | 156
Participants
  No Relief | 33 | 36 | 27
  Slight Relief | 83 | 83 | 46
  Moderate Relief | 115 | 111 | 58
  Marked Relief | 71 | 73 | 24
  Complete Relief | 12 | 11 | 1
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Superiority; p = 0.9915, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Test vs Placebo; Test type: Superiority; p = 0.0312, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Reference vs Placebo; Test type: Superiority; p = 0.0487, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: From first dose of randomized treatment until last dose plus 1-4 days (up to Day 15 + 3).
Description: Any signs or symptoms that occurs during randomized treatment period plus the 1-4 days post treatment.
Arm/Group | Test | Reference | Placebo
All-Cause Mortality (participants affected / at risk) | 0/317 | 0/320 | 0/158
Serious Adverse Events (participants affected / at risk) | 0/317 | 0/320 | 0/158
Other Adverse Events (participants affected / at risk) | 5/317 | 5/320 | 5/158
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=317) | Reference (N=320) | Placebo (N=158)
Headache (Nervous system disorders) | 5 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.